CLINICAL TRIAL: NCT04018066
Title: The Effect of Concord Grape Polyphenol-soy Protein Isolate Complex (GP-SPI) on Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Diana Roopchand, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2018002579
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Mechanisms, Defense
Keywords: gut microbiome; metabolome; dietary polyphenols; grape; nutrition

STUDY DESIGN:
Intervention Model Description: Longitudinal study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GP-SPI intervention (Experimental): 20 g of GP-SPI taken twice per day for 10 days
  Interventions: Dietary Supplement: GP-SPI

INTERVENTIONS:
Dietary Supplement: GP-SPI — grape polyphenol-soy protein isolate complex (GP-SPI)

SUMMARY:
The overall purpose of this study is to evaluate the effect of nutritional supplementation with a well-characterized preparation of Concord grape polyphenol-soy protein isolate (GP-SPI) on the composition of the gut microbiota.

DETAILED DESCRIPTION:
The proposed study will investigate how short-term supplementation with GP-SPI may modify the gut microbial community in healthy participants while monitoring liver and kidney function/health.

Significance:

Biochemical properties of the GP-SPI food ingredient are well-documented and GP-SPI and SPI supplements have been tested extensively in mice. The proposed study is a logical follow up to animal studies, which showed that compared to control mice fed a high-fat diet (HFD) supplemented with SPI alone, mice fed an isocaloric HFD supplemented with GP-SPI exhibited greater resistance to weight gain, adiposity, and glucose intolerance. These effects were accompanied by changes in murine gut microbiota composition, including increased abundance of the microbe Akkermansia muciniphila, associated with metabolic resilience. Similar gut microbiota changes were observed in lean mice fed low-fat diet (LFD) supplemented with GP-SPI.

The B-type proanthocyanidin (PAC) class of polyphenols contained in grape berries, especially skins and seeds, have been associated with health benefits; however, PACs are poorly absorbed and reach high concentration only in the colon raising questions about mechanism(s) of action. Prior studies showed that dietary PACs from grape and cranberry alter the gut microbiota in association with metabolic resilience. PACs are also biotransformed by gut bacteria to yield microbial metabolites (MMs) that may contribute to health benefits.

Research Design and Methods

Prospective participants will be recruited through flyers posted locally on Rutgers University campuses and sent to university email lists. Interested persons will be screened according to inclusion and exclusion criteria.

Enrolled subjects will begin the 17-day study.

Study Procedures

* Thirty subjects will be enrolled.
* Food List: Participants will maintain their usual diet except for a provided list of PAC-rich foods that they will be asked to abstain from for a 5-day wash-out period and during the 10-day intervention. The Food List is provided below. The goal is to have GP-SPI as the main/only source of PAC in the diet for the study period.
* Wash-out and SPI (Day -5 through -1): On day -5 (pre-baseline) before any supplementation, each subject will collect their fecal and urine sample. Each subject will then consume SPI twice a day (provided as pre-weighed packets of 20 g) during a 5-day wash-out period (days -5, -4, -3, -2, and -1). Subjects will be instructed to mix each packet of SPI in 250 mL of water or in a smoothie (recipe example below will be provided) using allowed foods as detailed in instructions and consume once in the morning before breakfast and once in the evening before dinner.
* Day 0: On the following day each subject will collect their baseline (day 0) stool and urine samples. They will have a blood sample drawn by a study nurse. Blood will be used for CMP test and prepared serum will be aliquoted and stored at -80 °C until processing for marker analysis and metabolomics. Analysis of day 0 samples should help isolate any effects due to SPI alone from subsequent samples collected during GP-SPI intervention. On day 0 subjects will drop off urine and stool samples at IFNH and collect GP-SPI packets. On Day 0 participants will also take a break from consuming SPI and will start GP-SPI supplementation on morning of Day 1.
* GP-SPI (Day 1 - 10): Each subject will receive twenty pre-weighed 20 g packets of GP-SPI. On day 1 subjects will be instructed to mix each packet of GP-SPI in 250 mL of water or in smoothie (recipe example will be provided, please see below) using allowed foods as detailed in instructions and consume the GP-SPI mix once in the morning before breakfast and once in the evening before dinner for 10 consecutive days.
* Subjects will be provided with a personal blender for smoothie preparation (value ~ $25) that they can keep.
* Digital food diary: Participants will be asked to take photos of all their food and drink (except water) including the study supplements with their personal mobile computing device (e.g. smart phone, iPad, or similar). Participants will be required to download the free mobile app WhatsApp to send photos with a brief description of the food items. Photos and food description may also be sent to an email address created for this study (food4microbes@sebs.rutgers.edu). The food diary must be kept over the 5-day SPI and wash-out period, day 0 (break day), the 10-day GP-SPI intervention period, and up until the final blood draw on day 11 (17 days total).
* Stool samples: Subjects will be provided with tubes containing 95% ethanol and/or tubes containing 50% glycerol (50% water) along with paper toilet accessories for easy self-collection of fecal samples; each participant will be instructed on use of stool collection materials. Fecal samples will be aliquoted and stored at -80 °C until extraction. Collection of fecal samples in 50% glycerol and immediate freezing will allow culturing of gut bacteria for in vitro experiments.
* Bristol stool scale form: Subjects will be provided with the Bristol stool scale (BSS) form and asked to complete it for stool samples they collect on days -5, 0, 2, 4, 6, 8, and 10 of the study. Stool consistency has been shown to strongly correlate with gut microbiota richness and composition, enterotypes, and bacterial growth rates. Subjects that report at least one bowel movement per day will be recruited for ease of compliance with study protocol. In addition, the BSS form contains an extra column to capture information about menstruation during time of sample collections as this variable could impact metabolite or bacteria profiles .
* Urine samples: Subjects will be provided with sterile collection containers for collection of urine samples on days 2, 4, 6, 8, 10 and asked to keep samples in 4 °C fridge until transport to the laboratory to maintain metabolite stability. Subjects will be asked to bring their samples to the laboratory as soon as possible, within 2-3 days of collection, for processing. Urine samples will be aliquoted and stored at -80 °C until processing for metabolomics studies.
* Blood sample: On day 11 subjects will have a final blood sample drawn. Blood will be used for CMP test and prepared serum will be aliquoted and stored at -80 °C until processing for marker analysis and metabolomics.

Samples will be used for a longitudinal, microbiome-wide association study (MWAS) to identify gut bacteria species/strains that are positively or negatively associated with GP-SPI supplementation. Metabolomics analysis will be performed on collected urine, fecal, and blood samples to identify/quantify known and unknown metabolites. Shotgun metagenomic sequencing will be performed on fecal samples to generate high quality draft genomes for species/strain level identification. These dynamic data sets will serve as input for the MWAS to correlate increasing/decreasing levels of gut bacterial species/strains to increasing/decreasing metabolites. These bacteria-metabolite associations will then be used to infer cause-effect relationships that can be further tested in vitro and in mouse models. We expect that successful completion of these studies will contribute to mechanistic explanations for how dietary polyphenols such as grape PACs alter the gut microbiota and resulting MM to promote metabolic health.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed based on a medical evaluation including a comprehensive metabolic panel (CMP) test with values in normal range, medical history and not presently taking any medication
2. Adults between 18 and 35 years
3. BMI 18.5 -29.9
4. Have at least one bowel movement per day
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. History/current cancer, rheumatoid arthritis immunologic, renal, hepatic, endocrine, neurologic or heart disease, hypertension, diabetes, GI dysfunction, or CMP test results showing values outside of normal range.
2. Cannot provide written informed consent.
3. Exposure to any experimental agent or procedure within 30 days of study.
4. Pregnancy or breast-feeding
5. Taking dietary supplements
6. Current smoker or have smoked within previous 6 months
7. Taking medications regularly (prescription, over the counter, supplements etc.)
8. Treated with antibiotics during the past 6 months
9. Have an allergy to soy or grapes

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Roopchand, PhD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers, The State University of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mezhibovsky E, Wu G, Wu Y, Ning Z, Bacalia K, Sadangi S, Patel R, Poulev A, Duran RM, Macor M, Coyle S, Lam YY, Raskin I, Figeys D, Zhao L, Roopchand DE. Grape polyphenols reduce fasting glucose and increase hyocholic acid in healthy humans: a meta-omics study. NPJ Sci Food. 2025 May 27;9(1):87. doi: 10.1038/s41538-025-00443-6. PMID 40425565
- See also: peer reviewed and published study — https://www.nature.com/articles/s41538-025-00443-6

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 participants were enrolled in the study based on inclusion/exclusion criteria. 4 participants withdrawn from the study, due to the following reasons: 3 started taking medications and 1 had scheduling conflicts. Of the remaining 30 participants that completed the study, 3 were excluded due to protocol deviations.
Groups:
- GP-SPI Intervention: Each participant consumed 20 g of soy protein isolate (SPI) twice per day for 5 days. After a one day break, participants then consumed 20 g of GP-SPI taken twice per day for 10 days. During the entire 17 day study period, participants abstained from an extensive list of PAC-rich foods.
  GP-SPI: grape polyphenol-soy protein isolate complex (GP-SPI)
Period: Overall Study
Arm/Group | GP-SPI Intervention
Started | 34 (34 participants were enrolled in the study)
Completed | 30 (30 participants completed the study protocol.)
Not Completed | 4
Not completed — participants started taking medications during the study period | 3
Not completed — participant dropped out due to schedule conflicts. | 1

BASELINE CHARACTERISTICS:
Population: 49 adults met initial inclusion/exclusion criteria. 11 people had CMP values outside normal ranges and 8 more people were excluded due to following reasons: 2 withdrew, 1 lost to follow up, 4 disqualified due to taking medication, 1 did not complete the study. 30 people completed study protocol, but 3 were excluded due to protocol deviations. 27 participants successfully completed the study protocol.
Arm/Group | GP-SPI Intervention
Number analyzed (Participants) | 27
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 21.7 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 27
Glucose [Mean (Standard Deviation); unit: mg/dL] | 88.78 (6.25)
Blood urea nitrogen [Mean (Standard Deviation); unit: mg/dL] | 12.81 (4.3)
Creatine [Mean (Standard Deviation); unit: mg/dL] | 0.76 (0.19)
Calcium [Mean (Standard Deviation); unit: mg/dL] | 9.82 (0.38)
Sodium [Mean (Standard Deviation); unit: mmol/L] | 142.7 (2.28)
Potassium [Mean (Standard Deviation); unit: mmol/L] | 4.83 (0.34)
Chloride [Mean (Standard Deviation); unit: mmol/L] | 103.4 (2.8)
Total carbon dioxide [Mean (Standard Deviation); unit: mmol/L] | 26.04 (1.72)
Anion gap [Mean (Standard Deviation); unit: meq/L] | 13.26 (2.19)
Protein [Mean (Standard Deviation); unit: g/dL] | 7.38 (0.37)
Albumin [Mean (Standard Deviation); unit: g/dL] | 4.83 (0.34)
Bilirubin total [Mean (Standard Deviation); unit: mg/dL] | 0.54 (0.26)
Alkaline phosphatase [Mean (Standard Deviation); unit: IU/L] | 68.56 (15.19)
Alkaline transaminase [Mean (Standard Deviation); unit: IU/L] | 21.26 (5.4)
Alanine transaminase [Mean (Standard Deviation); unit: IU/L] | 16.89 (7.44)

OUTCOME MEASURES:

1. Primary Outcome: Gut Microbiota Composition
Description: Evaluate the effect of nutritional supplementation with GP-SPI on gut microbiota composition by 16S rRNA amplicon sequencing and analysis
Time Frame: 16S rRNA amplicon sequencing will be performed on samples collected at baseline (before intervention, day -5), after 5 days of SPI supplementation (day 0), and after 10 days of GP-SPI supplementation (day 10). Total time frame is 17 days.
Population: All 27 participant samples were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of bacterial phyla
Arm/Group | GP-SPI Intervention
Number analyzed (Participants) | 27
percentage of bacterial phyla
  Firmicutes (day -5), % relative abundance | 58 (10)
  Bacteroidetes (day -5), % relative abundance | 30 (9.7)
  Verrucomicrobia (day -5), % relative abundance | 0.04 (0.1)
  Actinobacteria (day -5), % relative abundance | 7.3 (5.3)
  Proteobacteria (day -5), % relative abundance | 4 (2.9)
  Tenericutes (day -5), % relative abundance | 0.4 (0.1)
  Firmicutes (day 0), % relative abundance | 59.3 (6.9)
  Bacteroidetes (day 0), % relative abundance | 31.1 (8.06)
  Verrucomicrobia (day 0), % relative abundance | 0.04 (0.09)
  Actinobacteria (day 0), % relative abundance | 5.29 (3.7)
  Proteobacteria (day 0), % relative abundance | 3.66 (2.66)
  Tenericutes (day 0), % relative abundance | 0.009 (0.05)
  Firmicutes (day 10), % relative abundance | 54.3 (8.9)
  Bacteroidetes (day 10), % relative abundance | 33.44 (10.4)
  Verrucomicrobia (day 10), % relative abundance | 0.07 (0.13)
  Actinobacteria (day 10), % relative abundance | 8.1 (5.6)
  Proteobacteria (day 10), % relative abundance | 4.1 (2.6)
  Tenericutes (day 10), % relative abundance | 0.03 (0.1)

2. Secondary Outcome: Comprehensive Metabolic Panel (CMP) Blood Test (ALP, AST, ALT)
Description: Evaluate the effect of GP-SPI on kidney and liver health/function via CMP blood tests ALP, AST, ALT
Time Frame: Samples will be analyzed within one week of blood collection
Population: CMP data was measured for all 27 participants
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GP-SPI Intervention
Number analyzed (Participants) | 27
IU/L
  Alkaline phosphatase | 70.7 (16.79)
  Aspartate transaminase (IU/L) | 21.41 (5.6)
  Alkaline transaminase | 17.52 (8.59)

3. Secondary Outcome: Comprehensive Metabolic Panel (CMP) Blood Test (Glucose, Blood Urea Nitrogen, Creatine, Calcium, Bilirubin Total)
Description: Evaluate the effect of GP-SPI on kidney and liver health/function via CMP blood tests Measure glucose, blood urea nitrogen, creatine, calcium, bilirubin total
Time Frame: Samples will be analyzed within one week of blood collection
Population: CMP data was measured for all 27 participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GP-SPI Intervention
Number analyzed (Participants) | 27
mg/dL
  Glucose | 85.96 (6.79)
  Blood urea nitrogen | 14.81 (3.28)
  Creatine | 0.76 (0.18)
  Calcium | 9.64 (0.53)
  Bilirubin total | 0.54 (0.25)

4. Secondary Outcome: Comprehensive Metabolic Panel Blood Test (Anion Gap)
Description: The Anion gap was measured for all 27 participants. The anion gap is a calculation of the difference between the amounts of some negatively charged electrolytes (such as chloride and bicarbonate) and the amount of positively charged electrolytes (such as sodium) in blood. The anion gap reveals whether blood has an imbalance of electrolytes, i.e., blood is too acidic or too basic.
Time Frame: Samples will be analyzed within one week of blood collection
Population: CMP data was measured for all 27 participants
Measure: Mean (Standard Deviation); unit: meq/L
Arm/Group | GP-SPI Intervention
Number analyzed (Participants) | 27
meq/L | 14.41 (1.9)

5. Secondary Outcome: Comprehensive Metabolic Panel (CMP) Blood Test (Sodium, Potassium, Chloride, Total Carbon Dioxide)
Description: For all 27 participants CMP measured four electrolytes: sodium, potassium, chloride, total carbon dioxide. Electrolytes are minerals that carry an electric charge when they are dissolved in a liquid. These electrolytes in blood control nerve and muscle function and maintain the acid-base balance (pH balance) of blood and water balance.
  Sodium: Most sodium comes from food, and kidneys help regulate body's sodium levels.
  Potassium: Potassium comes from food and is present in all tissues of body. Bicarbonate: Bicarbonate indicates the amount of carbon dioxide (CO₂) in blood. Chloride: Chloride functions along with sodium, potassium and bicarbonate to control many processes in the body.
Time Frame: Samples will be analyzed within one week of blood collection
Population: CMP data was measured for all 27 participants
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | GP-SPI Intervention
Number analyzed (Participants) | 27
mmol/L
  Sodium | 142.2 (2.33)
  Potassium | 4.57 (0.43)
  Chloride | 102.3 (1.7)
  Total carbon dioxide | 25.51 (1.69)

6. Secondary Outcome: Comprehensive Metabolic Panel (CMP) Blood Test (Protein, Albumin)
Description: Evaluate the effect of GP-SPI on kidney and liver health/function via CMP blood tests
Time Frame: Samples will be analyzed within one week of blood collection
Population: CMP data was measured for all 27 participants
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | GP-SPI Intervention
Number analyzed (Participants) | 27
g/dL
  Protein | 7.37 (0.33)
  Albumin | 4.87 (0.29)

7. Secondary Outcome: Microbiome-wide Association Study
Description: Collect fecal, blood, and urine samples for a microbiome-wide association study (MWAS)
Time Frame: De-identified samples will be processed and analyzed after all subjects complete the study and within 1 year.
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Data Sharing
Description: Enter de-identified study results into microbiome and metabolome nationwide data sharing database
Time Frame: Data will be deposited no later than within 1 year of the completion of the funded project period for the parent award or upon acceptance of the data for publication, or public disclosure of a submitted patent application
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: 20 days
Description: An adverse event (AE) is any untoward medical occurrence in a subject during participation in the clinical study or with use of the experimental agent being studied. An adverse finding can include a sign, symptom, abnormal assessment (laboratory test value, vital signs, electrocardiogram finding, etc.), or any combination of these regardless of relationship to participation in the study.
Arm/Group | GP-SPI Intervention
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT04018066/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT04018066/ICF_001.pdf